CLINICAL TRIAL: NCT02090010
Title: Comparison of Two Needle Insertion Techniques on Success Rate and Complications During Subclavian Venous Catheterization: Seldinger vs. Modified Seldinger Technique
Brief Title: Subclavian Vein catheterization_Seldinger Vs Modified Seldinger
Acronym: MS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Pyoung Park, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Modified seldinger
Record Dates: First submitted 2014-03-16; First posted 2014-03-18 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-03

CONDITIONS: Brain Neoplasm; Intracranial Aneurysm; Cerebrovascular Moyamoya Disease
MeSH Terms: conditions — Brain Neoplasms; Intracranial Aneurysm; Moyamoya Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GroupC (Active Comparator): Group C means Control group which use Seldinger technique for subclavian catheterization. The aimed vessel(subclavian vein) is punctured with a sharp hollow needle, syringe is detached and guidewire is advanced through the lumen of the needle, and the needle is removed. After that catheter is passed over the guidewire into the vessel.
  Interventions: Procedure: Seldinger technique
- Group MS (Experimental): Group MS means experimental group which use modified Seldinger technique for subclavian catheterization. The aimed vessel is punctured with the needle that is covered with guiding sheath. After vessel is punctured, guiding sheath is instatntly slid over the needle into the vessel. The needle is removed, guidewire is advanced through the sheath, central catheter is placed into the vessel.
  Interventions: Procedure: Modified Seldinger technique

INTERVENTIONS:
Procedure: Seldinger technique — The aimed vessel(subclavian vein) is punctured with a sharp hollow needle, syringe is detached and guidewire is advanced through the lumen of the needle, and the needle is removed.
  After that catheter is passed over the guidewire into the vessel.
  Other Names: thin-wall needle technique
  Arms: GroupC
Procedure: Modified Seldinger technique — The aimed vessel is punctured with the needle that is covered with guiding sheath. After vessel is punctured, guiding sheath is instantly slid over the needle into the vessel. The needle is removed, guidewire is advanced through the sheath, central catheter is placed into the vessel.
  Other Names: guiding sheath-over-the-needle technique
  Arms: Group MS

SUMMARY:
Seldinger technique is a minimally invasive technique in which the practitioner accesses the target vessel with a small bore needle, then dilates to the size required for the catheter. Contrarily, modified Seldinger technique(guiding sheath-over-the-needle technique) use needle that is covered with guiding sheath.

Both technique is widely used in central venous catheterization, however, few researches have been investigated to compare success rate or complications of both methods.

DETAILED DESCRIPTION:
The major complications of central venous catheterization through subclavian vein, are unintended arterial puncture, pneumothorax, hemothorax, malposition of catheter etc,. We assume that using modified Seldinger technique (MST), guiding sheath is easily slid over the needle, providing stable route into the vessel lumen relatively.

We aimed to compare the Seldinger technique and modified Seldinger technique(MST) on success rate and complications during subclavian central venous catheterization in this prospective, randomized , controlled trials.

ELIGIBILITY:
Inclusion Criteria:

* patient scheduled for surgery under genearl anesthesia and subclavian vein central catheterization

Exclusion Criteria:

* Patient who does not agree to the study
* Inflammation or infection on catheterization site
* Contralateral diaphragmatic dysfunction
* Anatomic anomalies of subclavian artery or vein/clavicle
* Previous lung surgical history
* Patient who has ventriculoperitoneal shunt or chemoport on same side
* Patient who has pneumo/hemothorax or lung parenchymal disease

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Major complication rate of subclavian catheterization | intraoperative
  Compare main complication rates of subclavian catheterization including pnumothorax, hemothorax, arterial puncture, malposition of cathter.

SECONDARY OUTCOMES:
primary success rate of subclavian catheterization | intraoperative
  Check the number of attempts of needling, guidewire advance, and catheterization in both groups.
Total insertion time | From skin puctuation until confim the successful catheterization anticipated within 3min
  Check the total insertion time from skin puncture to confirm the successful catheterization via venous aspiration though catheter lumen.

CONTACTS AND LOCATIONS:
Overall Officials: Hee Pyung Park, MD PhD, Study Director — Professor; Eugene Kim, MD, Principal Investigator — Clinical Instuctor
Locations (1):
- Seoul National University of Hospital, Seoul, South Korea